CLINICAL TRIAL: NCT07267793
Title: Long-term Efficacy and Safety of CartiPRO Injection to Alleviate Knee Pain in Patients With Osteoarthritis and/or Diverse Cartilage Defects: a Multicenter, Single-blind, Randomized, Non-inferiority, Sponsor Initiated Trial
Brief Title: Long-Term Study of CartiPRO for Knee Pain Due to Osteoarthritis or Cartilage Damage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DALIM TISSEN Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DLTS_05
Record Dates: First submitted 2025-11-19; First posted 2025-12-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis; Knee Pain Arthritis; Cartilage Defects of the Knee; Knee Osteoarthritis; Degenerative Joint Disease of Knee
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Group applied with CartiPRO
  Interventions: Drug: Synovian®
- Control group (Active Comparator): Group applied with Synovian®
  Interventions: Device: CartiPRO

INTERVENTIONS:
Device: CartiPRO — Clinical subjects are enrolled after the investigator confirms eligibility, and subjects in the study group receive treatment Dalim Tissen's CartiPRO.
  Intra-articular medical device injection at baseline and Week 12; final assessment at Week 36.
  Arms: Control group
Drug: Synovian® — Clinical subjects are enrolled after the investigator confirms eligibility, and subjects in the study group receive treatment Synovian®. Intra-articular medical device injection at baseline and Week 12; final assessment at Week 36.
  Arms: Study Group

SUMMARY:
This clinical trial aims to evaluate and compare the efficacy and safety of CartiPRO, an approved intra-articular atelocollagen injection, versus Synovian injection for the relief of knee pain in patients with knee osteoarthritis. The investigational device is administered intra-articularly, with a second injection given 24 weeks after the first dose. Primary and secondary endpoints include changes in pain scores (VAS), functional assessments (WOMAC, SF-36), and safety evaluations over a 36-week period.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is the most common joint disorder, primarily caused by the destruction of articular cartilage. Symptoms typically include joint pain, stiffness, and muscle contraction. According to the World Health Organization, in 2013, an estimated 10-15% of adults over the age of 60 were affected by OA, significantly impacting their quality of life.

Collagen degradation is a key feature of cartilage damage in OA. Collagen-based injectable materials, such as atelocollagen, are being explored as potential therapeutic options to restore collagen and improve clinical outcomes. Unlike other injectable substances like hyaluronic acid or corticosteroids, collagen's stable triple helix structure and long half-life make it more resistant to enzymatic degradation, offering a potentially longer-lasting effect.

Despite this, long-term and repeated use data for atelocollagen injections in knee OA are limited both domestically and internationally. This study aims to provide robust clinical evidence on the efficacy and safety of repeated intra-articular atelocollagen injections for knee pain relief in patients with knee OA.

This is a randomized, single-blind, active-controlled study comparing CartiPRO with Synovian. Subjects with knee OA and symptomatic knee pain will receive the investigational device intra-articularly. A second dose will be administered at 24 weeks. The primary outcome is the change in 100-mm weight-bearing pain (WBP) VAS score at 12 weeks compared to baseline.

Secondary outcomes include VAS changes in WBP, resting pain (RP), motion pain (MP), and night pain (NP) at multiple time points, as well as changes in WOMAC and SF-36 scores. Long-term efficacy will be assessed after re-injection. Safety assessments include adverse events, local reactions, physical examination, vital signs, and laboratory tests.

Study Visits:

Visit 1: Screening Visit 2: First injection (baseline) Visit 3: 2 weeks after injection Visit 4: 4 weeks after injection Visit 5: 12 weeks after injection Visit 6: 24 weeks after injection (second dose) Visit 7: 36 weeks after first injection

ELIGIBILITY:
Inclusion Criteria

* Age 19 years and older
* Diagnosed with unilateral or bilateral knee osteoarthritis according to American College of Rheumatology (ACR) criteria, with at least 3 of the following 6 features:

  * Age ≥50 years
  * Morning stiffness <30 minutes
  * Crepitus on active motion
  * Bony tenderness
  * Bony enlargement
  * No palpable warmth
* Radiographic evidence of Kellgren-Lawrence grade I, II, or III osteoarthritis within 6 months prior to screening or at screening visit
* Weight-bearing pain Visual Analogue Scale (VAS) score ≥40 mm in at least one knee joint at screening
* Able to walk without assistive devices (walkers or canes), OR if using a walking aid routinely for past 6 months, able to continue using the same device throughout the study
* Able to understand and complete efficacy assessment questionnaires
* Willing and able to provide written informed consent

Exclusion Criteria

* Body Mass Index (BMI) ≥32 kg/m²
* Chronic inflammatory joint disease (e.g., rheumatoid arthritis)
* Inflammatory joint disease (e.g., septic arthritis)
* Secondary knee osteoarthritis due to ochronosis, hemochromatosis, or systemic disease
* Painful musculoskeletal conditions (e.g., Sudeck's atrophy, Paget's disease, herniated intervertebral disc)
* Polyarticular disease with severe osteoarthritis in other joints (e.g., hip) that may affect knee pain evaluation
* Radiographic evidence of definite loss of patellofemoral joint space
* Moderate to severe joint effusion confirmed by positive patellar tap test or equivalent
* History of myocardial infarction, congestive heart failure, other serious cardiac disease, or uncontrolled hypertension (≥140/90 mmHg despite treatment with ≥3 antihypertensive agents)
* History of autoimmune disease
* Active infection requiring parenteral antibiotics
* History of psychiatric disorder or epilepsy
* Cancer diagnosis within 5 years prior to screening
* Uncontrolled type 1 or type 2 diabetes mellitus (HbA1c >7%)
* Surgical procedures (including arthroscopy) on target knee within 1 year (surgery on contralateral knee or hip may be exclusionary if it could affect target knee assessment)
* Intra-articular corticosteroid injection into target knee within 12 weeks
* Systemic corticosteroid use within 4 weeks (topical and inhaled corticosteroids permitted)
* Surgery or radiation therapy to knee joint within 12 weeks, or not fully recovered from side effects
* Immunosuppressive therapy (e.g., Cyclosporine A, Azathioprine) within 6 weeks
* Intra-articular injections (e.g., hyaluronic acid) into knee joint within 6 months
* Prohibited concomitant medications within 2 weeks (unless washout period is adequate)
* Anticoagulants (e.g., warfarin, NOACs), antiplatelet agents (e.g., aspirin >100 mg/day, clopidogrel; low-dose aspirin ≤100 mg/day permitted), thrombolytic agents (e.g., urokinase, alteplase), or Vitamin E >1000 IU/day within 2 weeks (unless adequate washout)
* Habitual use (≥3 months) of psychoactive drugs or narcotic analgesics that may affect pain perception
* History of cell therapy or gene therapy to target joint
* Planned cell therapy or gene therapy to target joint
* Abnormal laboratory values at screening:
* ALT, AST, BUN, or serum creatinine >2× upper limit of normal
* Engaged in high-intensity aerobic or heavy anaerobic exercise that may affect the knee joint
* Dermatological disease at injection site or site deemed unsuitable for injection
* Ligament instability of Grade II or higher in target knee (Grade 0: none; Grade I: 0-5 mm; Grade II: 5-10 mm; Grade III: >10 mm)
* Known hypersensitivity to investigational product or its components
* Pregnant or breastfeeding women
* Women or men of childbearing potential unwilling to use acceptable contraception during study (acceptable methods: intrauterine device, tubal ligation, sterilization surgery, condom or diaphragm with spermicide, natural family planning)
* Participation in another clinical trial within 4 weeks
* Cognitive impairment or dementia preventing informed consent
* Any other condition that makes the subject unsuitable for study participation per investigator judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 100-mm Weight-Bearing Pain (WBP) Visual Analogue Scale (VAS) score (0-100 mm) | at week 12 after the first administration
  The change from baseline in Weight-Bearing Pain will be assessed using a 100-mm visual analogue scale ranging from 0 mm, no pain, to 100 mm, worst imaginable pain. Higher scores indicate more severe pain.

SECONDARY OUTCOMES:
Change from Baseline in Weight-Bearing Pain Visual Analogue Scale Score (0-100 mm) | at Weeks 2, 4, and 24 after the first administration
  The change from baseline in Weight-Bearing Pain will be assessed using a 100-mm visual analogue scale ranging from 0 mm, no pain, to 100 mm, worst imaginable pain. Higher scores indicate more severe pain.
Change from Baseline in Western Ontario and McMaster Universities Osteoarthritis Index Total and Subscale Scores | at Weeks 2, 4, 12, and 24 after the first administration
  The change from baseline in the Western Ontario and McMaster Universities Osteoarthritis Index will be assessed for the pain, stiffness, and physical function subscales, as well as the total score. Each item is rated from 0 to 4, where 0 indicates no symptoms and 4 indicates extreme symptoms. Subscale scores are calculated by summing item scores, and the total score is calculated as the sum of the subscale scores. Higher scores indicate worse symptoms and poorer function.
Change from Baseline in 36-Item Short Form Health Survey Domain Scores (SF-36) | at Weeks 2, 4, 12, and 24 after the first administration
  The change from baseline in the 36-Item Short Form Health Survey (SF-36) will be assessed using the eight domain scores: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Each domain score ranges from 0 to 100, where higher scores indicate better health status/quality of life.
Change from Baseline in Rest Pain Visual Analogue Scale Score (0-100 mm) | at Weeks 2, 4, 12, and 24 after the first administration
  The change from baseline in Rest Pain will be assessed using a 100-mm visual analogue scale ranging from 0 mm, no pain, to 100 mm, worst imaginable pain. Higher scores indicate worse pain.
Change from Baseline in Motion Pain Visual Analogue Scale Score (0-100 mm) | at Weeks 2, 4, 12, and 24 after the first administration
  The change from baseline in Motion Pain will be assessed using a 100-mm visual analogue scale ranging from 0 mm, no pain, to 100 mm, worst imaginable pain. Higher scores indicate more severe pain.
Change from Baseline in Night Pain Visual Analogue Scale Score (0-100 mm) | at Weeks 2, 4, 12, and 24 after the first administration
  The change from baseline in Night Pain will be assessed using a 100-mm visual analogue scale ranging from 0 mm, no pain, to 100 mm, worst imaginable pain. Higher scores indicate more severe pain.
Change from Week 24 (Re-administration) in Weight-Bearing Pain Visual Analogue Scale Score (0-100 mm) | at Week 36 (12 weeks after re-administration)
  The change from Week 24, defined as the time of re-administration, in Weight-Bearing Pain will be assessed using a 100-mm visual analogue scale ranging from 0 mm, no pain, to 100 mm, worst imaginable pain.Higher scores indicate worse pain.
Change from Week 24 (Re-administration) in Rest Pain Visual Analogue Scale Score (0-100 mm) | at Week 36 (12 weeks after re-administration)
  The change from Week 24, defined as the time of re-administration, in Rest Pain will be assessed using a 100-mm visual analogue scale ranging from 0 mm, no pain, to 100 mm, worst imaginable pain.Higher scores indicate worse pain.
Change from Week 24 (Re-administration) in Motion Pain Visual Analogue Scale Score (0-100 mm) | at Week 36 (12 weeks after re-administration)
  The change from Week 24, defined as the time of re-administration, in Motion Pain will be assessed using a 100-mm visual analogue scale ranging from 0 mm, no pain, to 100 mm, worst imaginable pain. Higher scores indicate more severe pain.
Change from Week 24 (Re-administration) in Night Pain Visual Analogue Scale Score (0-100 mm) | at Week 36 (12 weeks after re-administration)
  The change from Week 24, defined as the time of re-administration, in Night Pain will be assessed using a 100-mm visual analogue scale ranging from 0 mm, no pain, to 100 mm, worst imaginable pain. Higher scores indicate more severe pain.
Change from Week 24 (Re-administration) in Western Ontario and McMaster Universities Osteoarthritis Index Total and Subscale Scores | at Week 36 (12 weeks after re-administration)
  The change from Week 24, defined as the time of re-administration, in the Western Ontario and McMaster Universities Osteoarthritis Index will be assessed for the pain, stiffness, and physical function subscales, as well as the total score. Each item is rated from 0 to 4, where 0 indicates no symptoms and 4 indicates extreme symptoms. Subscale scores are calculated by summing item scores, and the total score is calculated as the sum of the subscale scores. Higher scores indicate worse symptoms and poorer function.
Change from Week 24 (Re-administration) in 36-Item Short Form Health Survey Domain Scores (SF-36) | at Week 36 (12 weeks after re-administration)
  The change from Week 24, defined as the time of re-administration, in the 36-Item Short Form Health Survey (SF-36) will be assessed using the eight domain scores: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Each domain score ranges from 0 to 100. Higher scores indicate better health status/quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yong In, Ph.D, Principal Investigator — The Catholic University of Korea
Locations (5):
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Bundang-gu
  - CHA Bundang Medical Center, Seoul, Bundang-gu
  - The Catholic University of Korea Eunpyeong St. Mary's Hospital, Seoul, Eunpyeong-gu
  - Gachon University Gil Hospital, Seoul, Namdong-gu
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, Seochogu

IPD SHARING:
Plan to Share IPD: Undecided
Undecided. The plan for sharing individual participant data has not yet been determined.